CLINICAL TRIAL: NCT04964167
Title: Indocyanine-green Mediated Photosensitizer VS Aloe Vera Gel: Adjunct Therapy to Scaling and Root Planing in Patients With Chronic Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Riyadh Elm University (Other)
Collaborators: Salah Abdalkreem Almohana (Unknown); Abdulmohsen Khalid Alanazi (Unknown); Abdulelah Khalid Alanazi (Unknown); Alhanouf Abdulkarem Almohana (Unknown)
Responsible Party: Principal Investigator, Zeeshan Qamar, Assistant Professor, Riyadh Elm University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FIRP/2021/94
Record Dates: First submitted 2021-06-28; First posted 2021-07-15 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Periodontitis; Periodontal Inflammation
MeSH Terms: conditions — Periodontitis | interventions — Plant Extracts

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Standard Root Planning) (Placebo Comparator)
  Interventions: Combination Product: Plant extract
- Group II (Standard Root Planning + Photodynamic Therapy) (Active Comparator)
  Interventions: Combination Product: Plant extract
- Group III (Standard Root Planning + Aloe Vera) (Experimental)
  Interventions: Combination Product: Plant extract

INTERVENTIONS:
Combination Product: Plant extract — Natural plant extract
  Other Names: Aloe Vera

SUMMARY:
For proving the potential of tropical medicaments on clinical parameters of periodontitis, a comprehensive assessment is required between therapeutic medicaments. The main aim of the study was to clinically evaluate and compare the efficacy of indocyanine green mediated photodynamic therapy (PDT) and aleo vera (AV) extract when used as an adjunct therapy to scaling and root planning (SRP) for treatment of chronic periodontitis.

One hundred and fifty patients included in this study were randomly distributed in three treatment groups Group I (SRP), Group II (SRP+PDT) and Group III (SRP+AV). Four clinical parameters plaque index (PI), bleeding on probing (BoP), periodontal (PD) pocket depth and clinical attachment level (CAL) were evaluated at three time points baseline, 3rd and 6th month respectively. Additionally the amount of three inflammatory cytokines IL-6, IL-8 and TNF- α in gingival crevicular fluid (GCF) was identified using enzyme linked immune-sorbent assay (ELISA) technique.

ELIGIBILITY:
Inclusion Criteria:

* age of ≥ 30 years;
* ≥ 20 natural teeth; and
* chronic-periodontitis (≥ 3 mm of CAL and PD pocket depth respectively on at least 30% of dental sites).

Exclusion Criteria:

* chronic systemic diseases;
* PD therapy during last 6 months;
* habitual use of chewable and non-chewable tobacco (smoking);
* alcohol consumers; or
* use of particular medications during last three months (steroidal and non-steroidal drugs/ anti-biotic/ anti-depressants)

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Clinically Evaluating the Effects of Topical Indocyanine-green Mediated Photosensitizer VS Aloe vera Gel: Adjunct therapy to Scaling and Root Planing in Patients with Chronic Periodontitis | 9 months
  Adjunct treatment regimens PDT and AV extract significantly helped in plummeting inflammation of PD tissue
IL-6 concentration in pg/ml | 6 months
  Identify the concentration of IL-6 in the gingival crevicular fluid
IL-8 concentration in pg/ml | 6 months
  Identify the concentration of IL-8 in the gingival crevicular fluid
TNF-α levels in pg/ml | 6 months
  Identify the concentration of TNF-α in the gingival crevicular fluid
Periodontal pocket depth in mm | 6 months
  Periodontal pocket depth
Clinical attachment loss in mm | 6 months
  Periodontal attachment loss

CONTACTS AND LOCATIONS:
Locations (2):
- Liaquat College of Medicine and Dentistry, Karachi, Pakistan
- Riyadh Elm University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No